CLINICAL TRIAL: NCT06580691
Title: Autologous Plasma Gel Injection Versus Polydioxanone Cog Threads Insertion for the Treatment of Atrophic Post-acne Scars: a Split-face
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sameh Sarsik (Other)
Responsible Party: Sponsor-Investigator, Sameh Sarsik, Lecturer, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 36264PR126/3/23
Record Dates: First submitted 2024-08-26; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Acne Vulgaris; Atrophic Acne Scar
Keywords: Acne vulgaris; Atrophic acne scars; Threads; Polydioxanone; Plasma gel
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Intervention Model Description: both male and female patients with atrophic acne scars
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Subcision plus Plasma gel (Active Comparator): The gel was injected into the scarred areas immediately after subcision.
  Interventions: Procedure: Subcision plus Plasma gel injection Vs Subcision plus Cog PDO threads
- Subcision plus Cog PDO threads (Active Comparator): Cog PDO threads were inserted using a blunt-tipped cannula in a "Z pattern" within the scarred areas, filling the pockets created by subcision.
  Interventions: Procedure: Subcision plus Plasma gel injection Vs Subcision plus Cog PDO threads

INTERVENTIONS:
Procedure: Subcision plus Plasma gel injection Vs Subcision plus Cog PDO threads — Plasma Gel: was injected into the scarred areas immediately after subcision. Thread Treatment: Cog PDO threads were inserted using a blunt-tipped cannula in a "Z pattern" within the scarred areas, filling the pockets created by subcision.

SUMMARY:
Both male and female patients, with atrophic acne scars

All patients underwent one session of subcision before receiving:

A: cog PDO threads on one side of the face (one session). B: plasma gel on the other side (one session). Primary outcomes: clinical improvements reported by physicians. Secondary out come: satisfaction levels of patients.

DETAILED DESCRIPTION:
The treatment area was prepared by anesthetizing the acne-scarred region with a 2% lidocaine injection mixed with 1/1000 adrenaline, administered at each entry point after sterilizing the area with povidone-iodine solution. Subcision was performed using an 18-G cannula needle inserted parallel to the skin surface. The skin was stretched while the needle was maneuvered along the scar margins on both sides of the face, creating a tunnel and releasing the scars from their bases. The procedure's endpoint was marked by a partial to complete loss of resistance in the treated area.

After subcision, patients underwent the following treatments:

Plasma Gel Therapy: One half of the face was assigned to the plasma gel therapy group. Plasma gel was prepared in two steps:

Platelet Poor Plasma (PPP) Preparation: Ten milliliters of venous blood were drawn from each patient and collected in sterile, anticoagulant-equipped vacuum tubes. The blood was centrifuged at 72 g for 15 minutes at room temperature, then the plasma layer was centrifuged again for 5 minutes at 1006 g to yield 6.5 ml of PPP and 0.5 ml of platelet-rich plasma (PRP).

Gel Formation: The PPP syringes were placed in a hot water bath (60-100°C) for 1 minute, then in a cold bath (8-0°C) for 1 minute to turn the plasma into a viscous gel. The gel was injected into the scarred areas immediately after subcision.

Thread Treatment: The other side of the face received PDO thread treatment. Cog PDO threads were inserted using a blunt-tipped cannula in a "Z pattern" within the scarred areas, filling the pockets created by subcision.

Randomization: Subcision was performed on both sides of the face, followed by either plasma gel injection or thread insertion. Patients were randomly assigned to either modality based on their patient number.

Assessment and Follow-up:

Assessments included standardized clinical photography, objective scar severity scoring, and patient-reported outcomes.

Clinical examination assessed the types and severity of acne scars using validated scales such as the Acne Scar Assessment Scale (ASAS), Goodman and Baron scale, ECCA grading scale, and Investigator Global Assessment (IGA) using a 5-point scale for improvement.

Patient satisfaction was measured using a 5-point scale from not satisfied to very satisfied. The Facial Acne Scar Quality of Life (FASQol) tool was used to assess the impact on patients' quality of life.

Photos were taken using a Samsung Galaxy S10 Plus smartphone with a 12 MP telephoto lens.

Participants were followed up at 4, 8, and 12 weeks post-treatment.

Outcome Measures:

The primary outcome measure was the change in scar severity scores from baseline to follow-up visits.

Secondary outcome measures included participant satisfaction scores, improvement in scar texture, and adverse events. Comparisons between treatment modalities were also made.

ELIGIBILITY:
Inclusion Criteria:

Patients over 18 years old, with atrophic acne scars on both sides of their faces of any severity.

Exclusion Criteria:

* patients with keloidal tendencies or bleeding disorders.
* Participants with a history of recent isotretinoin use within 3 months
* Patients who underwent any procedure for treatment of acne scars during the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Clinical improvement | after 3 month of the procedure
  The improvement was assessed using the Goodman and Baron scale.
Clinical improvement | after 3 month of the procedure
  The improvement was assessed using the ECCA grading scale.
Clinical improvement | after 3 month of the procedure
  The improvement was assessed using the physician global assessment.
Clinical improvement | after 3 month of the procedure
  The improvement was assessed using the FASQoL questionnaire to assess the effect on patients quality of life.

SECONDARY OUTCOMES:
Patients satisfaction. | 3 months from the procedure
  participant satisfaction score, improvement in scar texture.
Side effects of the procedures. | During 3 months from the procedure
  patients reporting of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Wael Saudi, MD, Principal Investigator — Misr University for Science and Technology
Locations (1):
- Department of Dermatology and Venereology, Faculty of Medicine, Tanta University, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No